CLINICAL TRIAL: NCT03415802
Title: Efficacy and Safety of Nab-Paclitaxel Plus S-1 in the First-line Treatment of Advanced Pancreatic Cancer: A Pilot Single Arm Phase II Study
Brief Title: Efficacy and Safety of Nab-Paclitaxel Plus S-1 in the First-line Treatment of Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aiping Zhou (Unknown)
Responsible Party: Sponsor-Investigator, Aiping Zhou, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-062
Record Dates: First submitted 2018-01-24; First posted 2018-01-30 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Advanced Pancreatic Cancer
Keywords: Nab-Paclitaxel; S-1; Advanced Pancreatic Cancer
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; S 1 (combination); Albumin-Bound Paclitaxel; Tegafur; gimeracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nab-paclitaxel Plus S-1 (Experimental): Nab-paclitaxel 120 mg/m2 (D1, D8, q3w) S-1 (40mg BID for body surface area<1.25 m2; 50mg BID for body surface area of 1.25-1.5m2; and 60mg BID for body surface area>1.5 m2; D1-14, q3w)
  Interventions: Drug: Nab-paclitaxel and S-1

INTERVENTIONS:
Drug: Nab-paclitaxel and S-1 — Nab-paclitaxel 120 mg/m2 (D1, D8, q3w) and S-1 (40mg BID for body surface area < 1.25 m2; 50mgBID for body surface area of 1.25-1.5 m2; and 60mg BID for body surface area >1.5 m2; D1-14, q3w)
  Other Names: Abraxane,Tegafur, Gimeracil and Oteracil Porassium

SUMMARY:
Pancreatic cancer is a common malignancy of digestive system with gradually increasing incidence, is the fourth and seventh leading cause of cancer-related mortality in the world (1) and China (2) according to the statistics in 2014. The vast majority of patients were confirmed as locally advanced or distantly metastatic disease at diagnosis with an estimated five-year survival rate of 4% (3) due to occlusive development and rapid progress. Advanced pancreatic cancer is characterized by poor prognosis.

DETAILED DESCRIPTION:
Gemcitabine has been approved as the standard chemotherapy for advanced pancreatic cancer since 1996, but the efficacy is extremely limited by a response rate of 6-8%, and median survival of 5.5-7 months. However, Gemcitabine-based combination treatments fail to transcend GEM monotherapy on overall survival, including GEM + 5-Fu [10], GEM + Oxaliplatin[11], and GEM + Irinotecan [12] and GEM + Cisplatin [13] (7-8) . Until 2011, Conroy et al.[15] reported that FOLFIRINOX solutions significantly improved ORR (31.6% vs 9%, P=0.0008), PFS (6.4 vs. 3.3 months, P<0.0001) and OS (11.1 vs. 6.8 months, P<0.001) than GEM single-agent, but the significant increase of grade 3/4 adverse reactions, to some extent, limited its wide application. Therefore, it is necessary to continue to explore effective and safe chemotherapy of advanced pancreatic cancer.

Nab-Paclitaxel was approved by FDA for advanced pancreatic cancer in September 2013. S-1 has demonstrated potential value in the treatment of advanced pancreatic cancer as a new compound oral 5-FU(4-5) and has been approved for pancreatic cancer treatment in Japan.

We conducted a single arm, prospective, phase II study in our center on the first-line treatment of advanced pancreatic cancer with nab-Paclitaxel and S-1 to investigate the efficacy and safety of the combination regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age, years: 18-75
* Histologically and cytologically confirmed advanced pancreatic cancer , inresectable, measurable lesions according to RECIST criteria; ECOG score of 0-1; life expectancy ≥12 weeks;
* Untreated; more than 6 months after the last adjuvant chemotherapy (does not include taxanes and S1);
* Laboratory examination within 14 days before entering the study should meet following requirements: ANC ≥ 1.5 x 10^9/L; PLT ≥ 100 x 10^9/L; Hb ≥ 90g/L (9g/dL); AST, ALT ≤ 2.5 x ULN (with no liver metastasis), ≤ 5 x ULN（with liver metastasis); creatinine ≤ 1.5 x ULN; TBIL ≤ 1.5 x ULN
* Both male and female subjects of potential fertility have to agree effective birth control during the entire study
* Informed consent

Exclusion Criteria:

* Concurrent other effective treatment (including radiotherapy)
* Resectable patients
* Allergy history to other drugs in the same class patients with pregnancy or lactation
* Known severe internal medical diseases
* Abnormal heart function or relevant history of myocardial infarction and severe arrhythmia
* Immunocompromised patients, such as HIV positive
* Uncontrollable mental illness
* Other conditions the researchers considered ineligible for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate（ORR） | 6 month
  CR+PR was defined as objective response rate (ORR)

SECONDARY OUTCOMES:
DCR | 6 month
  CR+PR+SD was defined as disease control rate (DCR)
PFS | 6 month
  From date of randomization until date of first documented PD, date of death
OS | 1 year
  From date of randomization until date of death
Safety profile: Adverse events of nab-Paclitaxel plus S-1 for advanced pancreatic cancer | 1 year
  Adverse events of nab-Paclitaxel plus S-1 for advanced pancreatic cancer

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, Doctor, Principal Investigator — National Cancer Center/Cancer Hospital, China
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese ACademy of Medical Sciences and Peking Union Medical College, Beijing, China